CLINICAL TRIAL: NCT06477276
Title: A Multicenter, Randomized, Controlled, Double-Blind Trial on the Efficacy and Safety of Amygdala Temporal Interference Stimulation for the Treatment of Depression.
Brief Title: Amygdala TIS for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Tianjin Anding Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, ZHANG CHENCHEHG, Clinical Neuroscience Center Deputy Director, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024LLSD160-001
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
Keywords: Deep Brain Stimulation; Non-invasive; TI; Amygdala; Temporal Interference
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amygdala TI (Experimental): 5 sessions will be delivered in 3 weeks
  Interventions: Device: Nervio-X
- Controlled TI (Sham Comparator): 5 sessions will be delivered in 3 weeks
  Interventions: Device: Nervio-X

INTERVENTIONS:
Device: Nervio-X — An 8-channel TIS device developed by NEURODOME Corporation.

SUMMARY:
The current investigation employs a directed neuromodulation technique, specifically targeting the right amygdala, to ascertain its therapeutic efficacy in managing depressive episodes. The intervention's safety and efficacy will be evaluated using an assessment incorporating depressive symptomatology, cognitive abilities, and daily functions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged between 18 and 65, with no gender restrictions;
* A diagnosis of depression made by the study physician based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
* HAMD-17 score of 17 or higher;
* Participants must not have changed their antidepressant medication regimen from 30 days prior to signing the informed consent form through the duration of the experiment;
* Eligible individuals or their authorized representatives must demonstrate, as assessed by the study physician, a comprehensive understanding of the study's objectives and procedures, be capable of adhering to the requirements set forth in the study protocol and provide their signature on the informed consent form.

Exclusion Criteria:

* Eligible participants must not have a history of psychiatric disorders such as schizophrenia, as judged by the investigator, which may impact the evaluation of the study's efficacy;
* Participants must not have a history of seizures or prior episodes of epilepsy;
* The presence of metallic foreign objects within the cranial structure or metallic cardiac implants;
* Participants must not have a diagnosis of organic brain disease nor a history of significant cranial trauma or neurosurgical intervention;
* Participants received electroconvulsive therapy or other physical therapies (such as transcranial magnetic stimulation therapy);
* The researcher evaluated the individual's mental state and determined it to present a significant risk of suicidal ideation or behavior;
* Pregnant or breastfeeding;
* Participants who are concurrently engaged in other clinical interventional trials;
* Participants presenting with other circumstances that the investigator deems unsuitable for the intervention being studied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self-Report (16-item version) | 4 weeks

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (17-item version) | Baseline, 1 week, 4 weeks and 8 weeks
Quick Inventory of Depressive Symptomatology - Self-Report (16-item version) | Baseline, 1 week and 8 weeks
Snaith-Hamilton Pleasure Scale | Baseline, 1 week, 4 weeks and 8 weeks
  The SHAPS is a questionnaire that used to measure the severity of anhedonia, a common symptom in various mental health conditions.
Hamilton Anxiety Rating Scale | Baseline, 4 weeks and 8 weeks
Pittsburgh Sleep Quality Index | Baseline, 4 weeks and 8 weeks
36-Item Short Form Health Survey | Baseline and 8 weeks
World Health Organization Quality of Life Assessment - Brief Version | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, MD PhD, Principal Investigator — Ruijin Hospital
Locations (3):
- China (3):
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai
  - Tianjin Anding Hospital (Mental Health Center of Tianjin Medical University), Tianjin

IPD SHARING:
Plan to Share IPD: No